CLINICAL TRIAL: NCT07355257
Title: Safety and Efficacy of Telitacicept in Inflammatory Myopathies
Brief Title: TELITACICEPT IN INFLAMMATORY MYOPATHIES(TELITACICEPT-IM)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professer, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-362
Record Dates: First submitted 2026-01-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Myopathy
MeSH Terms: conditions — Myositis | interventions — telitacicept

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Treatment group (Experimental)
  Interventions: Drug: Telitacicept 240mg

INTERVENTIONS:
Drug: Telitacicept 240mg — On the basis of the original foundational medication regimen, add Telitacicept 240mg administered via subcutaneous injection once a week for a total of 12 weeks.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of Telitacicept in the treatment of inflammatory myopathy in patients with inflammatory diseases. The main question it aims to answer is: the safety and effectiveness of Telitacicept in treating inflammatory myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 70 years.
* Patient has a confirmed diagnosis of inflammatory myopathy, meeting the 2017 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for idiopathic inflammatory myopathies.
* Inadequate response or intolerance to glucocorticoids and/or at least one immunosuppressant.
* The patient or their legal guardian provides written informed consent.

Exclusion Criteria:

* Female patients who are pregnant, breastfeeding, or planning a pregnancy during the trial period.
* Patients with active infections, such as herpes zoster, HIV, active tuberculosis, active hepatitis, HBsAg-positive patients, or HCV antibody-positive patients.
* Patients with positive test results indicating COVID-19 infection within 1 month prior to baseline.
* Patients with a history of or currently diagnosed malignancy.
* Patients with significant cardiovascular diseases (including severe arrhythmia), hepatic, renal, respiratory, endocrine, or hematological disorders, or any other medical condition that, in the investigator's judgment, would interfere with participation in the study or require hospitalization during the trial.
* Patients who have received intravenous immunoglobulin (IVIG) or plasmapheresis within 1 month prior to baseline.
* Patients who have received other targeted biologic therapies, such as rituximab, eculizumab, tocilizumab, etc., within 3 months prior to baseline.
* Patients who have received any live vaccine within 3 months prior to baseline or plan to receive any vaccine during the study period.
* Patients with a known allergy to human-derived biologics.
* Patients currently participating in another clinical trial.
* Patients deemed unsuitable for participation by the investigator for other reasons (e.g., severe psychiatric disorders).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) Score | From enrollment to the end of treatment at 12 weeks